CLINICAL TRIAL: NCT06142526
Title: A Randomized and Single-blinded Pilot Study to Evaluate the Safety and Effectiveness of DividPro Film in Open Abdominal Surgery
Brief Title: A Safety and Effectiveness Study of DividPro Film in Open Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Industrial Technology Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITRIDP20220510
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Open Abdominal Surgery; Abdominal Adhesion
Keywords: adhesion barrier; abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): DividPro film implantation right before the closure of surgical incision wound
  Interventions: Device: DividPro film
- control group (No Intervention): Only standard care without any anti-adhesion related products.

INTERVENTIONS:
Device: DividPro film — DividPro Film is a sterile biodegradable translucent film that served as a physical barrier for preventing the adhesion between two adjacent layers of tissue in wound healing process.
  Arms: treatment group

SUMMARY:
Abdominal adhesions frequently occur after surgery and may be one of the main reasons to cause discomfort, pain and related bowel movement symptoms. The goal of this clinical trial is to evaluate the safety of DividPro film and its potential effectiveness for reducing the incidence of abdominal adhesion. Treatment group will have DividPro film implantation right before the closure of surgical incision wound. Control group will have standard care without any anti-adhesion related products. In addition to adverse event assessment and safety lab tests, participants will accept abdominal ultrasound and quality of life questionnaire at each visit for effectiveness evaluation.

DETAILED DESCRIPTION:
Adhesion may occur due to the excessive production of fibrous tissue during the process of wound healing. Abdominal adhesion could play a role on intestine obstruction which will lead to lack of blood flow to the blocked part of the intestine or peritonitis. Improving surgical skills, cleaning wound before closure or using physical barrier between the incision site and abdominal wall can lower the incidence of abdominal adhesion.

In this study, participant who meets the eligibility criteria will be enrolled and randomized to either the treatment or control group. During the surgery period, subject will have the DividPro film implantation or only the standard care procedure right before the closure of the surgical wound. Participants will be instructed to return for visits on day 7, month 1, 3, 6 and 12. Adverse event, clinical laboratory test, vital sign and physical examination will be tested and recorded during the course of the study as the items of safety assessment. In addition, symptom related to tissue adhesion, visceral sliding test and quality of life questionnaire will also be assessed as the parameters of efficacy at the predetermined time points throughout the study .

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study specific procedure is performed.
2. Ages of 20-70 years old on the day of consent.
3. Subject who is diagnosed with a liver, gallbladder, pancreas and upper/lower gastrointestinal disorder.
4. Subject who is scheduled to accept an open abdominal operation involving liver, gallbladder, pancreas, stomach, spleen, intestine or female pelvic organ.
5. The Investigational product can be implanted appropriately between the surgical wound and operated organ and is able to cover the entire wound area.

Exclusion Criteria:

1. Subject who is hypersensitive to the ingredient of DividPro film [Poly (DL-lactide)]
2. Subject who is concurrently participating in another clinical trial with a drug or a device.
3. Subject who has taken Immunosuppressive drugs/agents long-term or taken NSAIDs within 7 days before trial's operation.
4. Subject who has participated in a clinical trial with a drug or a device within 30 days prior to this study.
5. Subject who has received or is expected to receive any other product or technique belonging to the group of adhesion reduction devices or other products, meshes, or other types of implants in the abdominal cavity within 30 days prior to or during enrollment.
6. Subject who has had hernia mesh placed under the abdominal wall.
7. Subject with peritonitis.
8. Subject with hematological, neurological or immune critical illness.
9. Subject who has malnutrition, uncontrolled diabetes or any other conditions that the investigator considers might not be suitable for enrollment to the study.
10. Subject with other potential infections.
11. Subject with BMI≧40.
12. Female subject who is lactating or pregnant.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events and the incidence of both respectively | from baseline to day 7, and 1, 3, 6 and 12 month
Incidence of adhesion by using visceral sliding test | from baseline to 3 month

SECONDARY OUTCOMES:
Safety profiles assessment by evaluating the changes in physical examination | from baseline to day 7, and 1, 3, 6 and 12 month
Safety profiles assessment by evaluating the changes in laboratory data | from baseline to day 7, and 1, 3, 6 and 12 month
Safety profiles assessment by evaluating the changes in vital signs | from baseline to day 7, and 1, 3, 6 and 12 month
Incidence of adhesion by using visceral sliding test | from baseline to day 7, and 1, 6 and 12 month
Changes in the score of Small Bowel Obstruction Questionnaire | from baseline to day 7, and 1, 3, 6 and 12 month
  The questionnaire includes measurements for the impact of small bowel obstruction on the patients' quality of life in respect to diet, pain, gastrointestinal symptoms and daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Ming Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan